CLINICAL TRIAL: NCT03468374
Title: Role of Sentinel Lymph Node Identification in Patients With Breast Cancer Using SPECT/CT
Brief Title: Sentinel Lymph Node Identification in Patients With Breast Cancer Using SPECT/CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Raghda Hassan Mohamed Farweiz, Assiut Medical School Ethical Review Board, Assiut University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: SLN SPECT
Record Dates: First submitted 2018-03-04; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-02

CONDITIONS: Early-stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lymphoscintigraphy; Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphoscintigraphy (Active Comparator): Nuclear Medicine diagnostic device using radioactive material
  Interventions: Device: lymphoscintigraphy
- Single Photon Emission Tomography (Active Comparator): Nuclear Medicine diagnostic device using fusion technique between SPECT and CT
  Interventions: Device: Single Photon Emission Tomography

INTERVENTIONS:
Device: lymphoscintigraphy — Nuclear Medicine diagnostic device using radioactive material
  Arms: Lymphoscintigraphy
Device: Single Photon Emission Tomography — Nuclear Medicine diagnostic device using fusion technique between SPECT and CT
  Arms: Single Photon Emission Tomography

SUMMARY:
Role of SPECT/CT in detection of sentinel lymph node in patients with breast cancer that is in early stage with small mass with no nodal or distant metastasis using radioactive material nannocolloid that can change surgical approach

DETAILED DESCRIPTION:
The status of axillary lymph node involvement is the best prognostic factor in patients with early stage breast cancer. In the past; removal of all of the axillary lymph nodes (axillary lymph node dissection, ALND) was often the preferred method of treatment.

ALND, however, has significant short- and long-term morbidity, the most significant being lymphoedema. With the trend towards earlier detection and presentation of breast cancer, most patients do not have lymphatic metastases at diagnosis.

In these patients, ALND is purely a diagnostic procedure, with no therapeutic benefit; besides the widespread use of breast conserving surgery, the staging procedure carries greater morbidity than the therapeutic procedure of the primary cancer.

Sentinel lymph nodes (SLNs) are defined as the first lymph nodes in a tumor bed that receive lymphatic drainage directly from the primary tumor; accordingly these nodes are most likely to harbor metastasizing cancer cells along the path of lymph drainage of tumor tissues, if lymphatic metastasis does occur.

SLN biopsy (SLNB) has been demonstrated to be an ideal option to accurately stage axillary nodal involvement in breast cancer; it is a minimally invasive technique for lymphatic staging. The accurate detection of the SLN is paramount for the success of the procedure.

SLNB in patients with clinically node-negative breast cancer is a valuable procedure for nodal staging ,treatment selection guiding, and often spares patients from the potentially devastating side effects of ALND such as lymphedema while maintaining the curative effect of surgery.

Although being an important element in identification of SLNs; interpretation of planar lymphoscintigraphy is hindered by the absence of anatomical landmarks in the scintigraphic image.

Single photon emission computed tomography coupled with computed tomography (SPECT/CT) was introduced in lymphatic mapping with the goal to show more SLNs and to show them more clearly than is possible with planar lymphoscintigraphy to improve nodal staging.

Besides providing functional scintigraphic information, it provides accurate anatomical localization. This advantage facilitates surgical exploration.

SPECT/CT can detect additional nodes not visualized on planar images and is especially useful in visualization of SLN outside the axilla or nodes close to the injection site.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18≤ years' old, female gender.
* Patients with histopathologically proven breast cancer.
* Patients with early stage and invasive breast cancer stage T1 with mass no more than 2 cm in greatest dimension or stage T2 with mass more than 2 cm but no more than 5 cm in greatest dimension with no clinical evidence of axillary lymph node metastasis(N0) and no remote metastasis (M0).

Exclusion Criteria:

* Patients with LABC, multifocal breast cancer or distant metastasis.
* Clinical, histological or radiological evidence of regional nodal metastasis.
* Prior major breast or axillary operations that could interfere with lymphatic drainage.
* Pregnancy.
* Inability to sign informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Role of SPECT/CT in sentinel lymph node detection in breast cancer | 3 years
  Early detection of sentinel lymph node in patients with breast cancer using SPECT/CT by radioactive material nanocolloid to change surgical approach

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Samphao S, Eremin JM, El-Sheemy M, Eremin O. Management of the axilla in women with breast cancer: current clinical practice and a new selective targeted approach. Ann Surg Oncol. 2008 May;15(5):1282-96. doi: 10.1245/s10434-008-9863-8. Epub 2008 Mar 11. PMID 18330650
- [Background] Giuliano AE, Kirgan DM, Guenther JM, Morton DL. Lymphatic mapping and sentinel lymphadenectomy for breast cancer. Ann Surg. 1994 Sep;220(3):391-8; discussion 398-401. doi: 10.1097/00000658-199409000-00015. PMID 8092905
- [Background] Kim T, Giuliano AE, Lyman GH. Lymphatic mapping and sentinel lymph node biopsy in early-stage breast carcinoma: a metaanalysis. Cancer. 2006 Jan 1;106(1):4-16. doi: 10.1002/cncr.21568. PMID 16329134
- [Background] Cheng G, Kurita S, Torigian DA, Alavi A. Current status of sentinel lymph-node biopsy in patients with breast cancer. Eur J Nucl Med Mol Imaging. 2011 Mar;38(3):562-75. doi: 10.1007/s00259-010-1577-z. Epub 2010 Aug 11. PMID 20700739
- [Background] Somasundaram SK, Chicken DW, Keshtgar MR. Detection of the sentinel lymph node in breast cancer. Br Med Bull. 2007;84:117-31. doi: 10.1093/bmb/ldm032. Epub 2008 Jan 3. PMID 18174216
- [Background] Sadeghi R, Forghani MN, Memar B, Abdollahi A, Zakavi SR, Mashhadi MT, Raziee HR, Tavassoli A, Kakhki VR. Comparison of pre-operative lymphoscintigraphy with inter-operative gamma probe and dye technique regarding the number of detected sentinel lymph nodes. Hell J Nucl Med. 2009 Jan-Apr;12(1):30-2. PMID 19330179
- [Background] Hubalewska-Dydejczyk A, Sowa-Staszczak A, Huszno B. Current application of sentinel lymph node lymphoscintigraphy to detect various cancer metastases. Hell J Nucl Med. 2006 Jan-Apr;9(1):5-9. PMID 16617387